CLINICAL TRIAL: NCT05741112
Title: The Long COVID-19 Wearable Device Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Julia Moore Vogel, Director, Scripps Translational Science Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LCWS 001
Record Dates: First submitted 2023-02-17; First posted 2023-02-23 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Long COVID; Postural Orthostatic Tachycardia Syndrome; Dysautonomia; Myalgic Encephalomyelitis; Chronic Fatigue Syndrome; Long Covid19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Postural Orthostatic Tachycardia Syndrome; Autonomic Nervous System Diseases; Fatigue Syndrome, Chronic | interventions — Wearable Electronic Devices

STUDY DESIGN:
Intervention Model Description: All participants will have a diagnosis of Long COVID-19, Chronic Fatigue Syndrome or Postural Orthostatic Tachycardia Syndrome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control: study provided wearables (Other): Following consent and the completion of the baseline assessments the control group will receive basic education on symptom management. At the 3 month timepoint they will be prompted to order their device and receive enhanced education that will provide information on how wearable devices can be used to monitor and manage symptoms.
  Interventions: Device: Wearable device
- Treatment: study provided wearables (Other): Following consent and the completion of the baseline assessments the treatment group will be prompted to order their device and receive basic education on symptom management along with the enhanced education on wearable devices.
  Interventions: Device: Wearable device
- Control: self provided wearables (Other): Following consent and the completion of the baseline assessments the control group will receive basic education on symptom management. At the 3 month timepoint they will be receive enhanced education that will provide information on how wearable devices can be used to monitor and manage symptoms.
  Interventions: Device: Wearable device
- Treatment: self provided wearables (Other): Following consent and the completion of the baseline assessments the treatment group will receive basic education on symptom management along with the enhanced education on wearable devices.
  Interventions: Device: Wearable device

INTERVENTIONS:
Device: Wearable device — The treatment group will receive their wearable device and the enhanced education at the start of the study. Their outcomes will be compared with the control group who will receive at 3 months.
  Other Names: Educational materials

SUMMARY:
To further characterize Long COVID-19 by collecting data from individuals who already own wearable devices or are provided with a wearable device along with basic and enhanced educational materials to determine if both can improve Long COVID-19 symptom management and post-exertional malaise.

DETAILED DESCRIPTION:
This study will have two components:

One study group will consist of up to 100,000 individuals who own wearable devices and are willing to share their data. These participants will be randomized and will receive educational materials. The investigators will study these dynamic wearable data along with participant survey responses that focus on diagnoses, symptoms, and quality of life to improve disease characterization and understanding of differences within and between individuals.

The other group in the randomized trial will participants who do not already own a wearable device. The study will distribute wearable devices and pacing educational materials to 500 individuals who do not already own them and experience post-exertional malaise, or the worsening of symptoms following exertion.

The investigators hypothesize that access to personalized information from a wearable device will enable participants to reduce post-exertional malaise. The investigators will include up to 25% individuals whose post-exertional malaise is caused by a condition other than Long COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years old.
* Has a self/and or physician diagnosis of:
* Long COVID (based on the WHO working definition),
* ME/CFS (myalgic encephalomyelitis / chronic fatigue syndrome, self-diagnosis based on IOM criteria), and/or
* POTS (Postural Orthostatic Tachycardia Syndrome).
* Is interested in tools to manage ME/CFS, POTS, and/or Long COVID symptoms.
* Owns a wearable device they are willing to use for this study or does not own a device and agrees to utilize a study-provided one.
* Agrees to wear the device throughout the study period, share the data with the study, and sync data at least weekly.
* Has access to a smartphone or tablet to enable syncing wearable data and viewing device feedback.
* Agrees to disclose involvement in other ME/CFS, POTS, and/or Long COVID interventions such as medical treatment, self-management, and other interventional studies.
* Agrees to complete at least 75% of the study surveys.

Exclusion Criteria:

* As long as they meet inclusion there is no exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100500 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary Objective 1:Assess the effect of study-provided devices and enhanced educational materials to manage Long COVID-19 symptom severity, compared to general educational materials alone using data from participants survey responses. | 3 months
  Will measure relapse symptom frequency, symptom severity, pain, quality of life and overall health through the analysis and measurement of change in the weekly survey responses.
Primary Objective 2: Collate a unique longitudinal dataset combining patients' demographics, symptoms, symptom severity, quality of life, and sensor data including sleep, activity, heart rate, heart rate variability, and Body Battery. | 12 months
  Will measure relapse symptom frequency, symptom severity, pain, quality of life and overall health through the analysis and measurement of change from the baseline survey to the quarterly survey.

SECONDARY OUTCOMES:
Secondary Objective: Assess the longitudinal impact of sustained use of the study-provided devices and enhanced educational materials on symptom severity. | 12 months
  Conduct within-subject comparisons on the primary and secondary endpoints listed above but such that the investigators are assessing the change between the baseline measurement at month zero and that of the quarterly survey nine months after the distribution of the device and/or enhanced education materials.

OTHER OUTCOMES:
Exploratory Objective: Assess whether individuals who enroll in the study with their own wrist-worn wearable device and receive educational materials see a decrease in symptom severity and whether this differs by device brand and/or feature. | 12 months
  Cross-referencing heart rate patterns with participant-provided symptoms and diagnoses to identify correlations; identify underlying signals in surveys and/or wearable data that may help differentiate those who will recover within six months from those who will not recover for years; identify correlates with which individuals experience worsening symptoms over time, such as whether consistent reduced heart rate variability affects long-term symptoms as it does short-term symptoms. The self-provided wearable cohort can share data from the complete history of their wearable device (and in some cases the history from their ownership of a device of the same brand), therefore the investigators can also conduct within-subject analysis for those that were using a wearable device prior to their COVID-19 infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Scripps Research, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators may share the coded study data with researchers outside of Scripps Research. Before doing so, they will ensure that nothing in the data can identify the participant directly.